CLINICAL TRIAL: NCT07029646
Title: Comparative Research on the Accuracy of Margin Interpretation in Breast-Conserving Surgery for Breast Cancer: Cell Microscopic Imaging and Standard Frozen Pathology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, zhaoqingfan, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-P37
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Breast-Conserving Surgery; Breast Carcinoma; Margins in the Specimen
Keywords: Breast-Conserving Surgery; Breast Cancer; Margins; microscope
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): Use of EndoScell™ intraoperative handheld microscope
  Interventions: Device: EndoScell™ intraoperative handheld microscope
- FS group (No Intervention): without the use of EndoScell™ intraoperative handheld microscope

INTERVENTIONS:
Device: EndoScell™ intraoperative handheld microscope — The research instrument used is the EndoScell™ intraoperative handheld microscope, which employs the principle of epifluorescence. It is a miniaturized microscope that reduces the size of a traditional large optical microscope by approximately a thousand times. It is the world's first handheld micrometer-level intraoperative real-time cell imaging probe microscope. This microscope is equipped with high-definition, real-time, anti-shake, and full-coverage scanning features. It can rapidly investigate the structure and cell morphology of tissues in real-time.
  Arms: ES group

SUMMARY:
The goal of this clinical trial is to assess whether cell microscopic imaging can accurately determine the tumor-free status of surgical margins in breast cancer patients undergoing breast-conserving surgery. This study involves female patients aged 18-70 years with breast cancer who are candidates for breast-conserving surgery. The main question it aims to answer is:

- Can cell microscopic imaging provide accurate intraoperative assessment of surgical margins compared to standard frozen pathology?

Researchers will compare the results of cell microscopic imaging to those of standard frozen pathology and paraffin pathology to see if the new imaging technology can effectively and quickly determine whether surgical margins are free of cancer cells.

Participants will:

* Undergo breast-conserving surgery with standard pathological assessments.
* Have their surgical margins evaluated using cell microscopic imaging during the operation.
* Be monitored for postoperative recovery at regular intervals (2 weeks, 3 months, 6 months, and 12 months) after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old;
* Clinical or imaging showed a single lesion with no evidence of distant metastasis;
* No invasion of the skin, subcutaneous tissue, pectoralis major muscle, and nipple-areola complex;
* Breast cancer patients who are willing to undergo breast-conserving surgery;
* Subjects voluntarily signed the informed consent form.

Exclusion Criteria:

* Allergic constitution;
* Chest wall or skin invasion, locally advanced breast cancer;
* Extensive axillary lymph node metastasis (stage ⅢB and above);
* Patients with severe complications (such as organ dysfunction, immunodeficiency) and poor general condition;
* Unable to accept general anesthesia or surgical treatment;
* Participating in other clinical studies that may affect this trial;
* Patients who cannot send frozen pathology and paraffin pathology specimens for examination during surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Within 7 days after the operation
  Compare the results of cell microscopic imaging to those of standard frozen section and paraffin section pathology to determine the accuracy and potential advantages of the new imaging technology in real-time intraoperative assessment of surgical margins